CLINICAL TRIAL: NCT03761121
Title: Developing Fast Pediatric Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ellen Grant, Principal Investigator, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18-325; R01EB020613 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-12-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Low-grade Gliomas
Keywords: Neuro Oncology

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary Testing Group (Experimental): * This scan is in the same imaging session as the participant's scheduled clinical MRI and is no longer 15 minutes
  * Wave-CAIPI will be use to enable a 40-60 s acquisition per contrast at 0.9-mm isotropic resolution
  * Wave-CAIPI will be used to acquire a 4-echo GE-SE time-series at 1.5-mm isotropic resolution
  Interventions: Other: Wave-CAIPI
- Software Testing Group (Experimental): * Participants will receive hour research-only scan
  * Wave-CAIPI will be use to enable a 40-60 s acquisition per contrast at 0.9-mm isotropic resolution
  * Wave-CAIPI will be used to acquire a 4-echo GE-SE time-series at 1.5-mm isotropic resolution
  Interventions: Other: Wave-CAIPI

INTERVENTIONS:
Other: Wave-CAIPI — "wave-CAIPI" technology, a data acquisition / reconstruction scheme designed to optimally exploit available information in modern multi-channel receivers and in multi-contrast/time-series data for improved image encoding

SUMMARY:
This research study is evaluating the investigational software for magnetic resonance imaging (MRI) systems and techniques to process magnetic resonance (MR) images

DETAILED DESCRIPTION:
The purpose of the study is to develop new technologies for MRI systems. The new technologies should improve MRI capabilities in terms of how sensitive, specific, and efficient they are. The overall goal is to get better measurements of the brain tumor tissue(s).

In this research study, the investigators want to learn more about investigational software and about techniques to process MR images. The testing of investigational software will allow the investigators to improve the image quality. As part of the testing process, the investigators will collect more MR images of the brain, and improve current image reconstruction methods. This will allow a more precise analysis of MR images and potentially better assessment of the brain tumor tissue volume.

ELIGIBILITY:
Inclusion Criteria:

* Infants, children and adults who have been diagnosed with Low Grade Glioma
* Healthy volunteers - Children from age 0 to adults with no upper age limit or;
* Diagnosed with LGG and being treated at DFCI;

Exclusion Criteria:

* Electrical implants such as cardiac pacemakers or perfusion pumps;
* Ferromagnetic implants such as aneurysm clips, surgical clips, prosthesis, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants;
* Ferromagnetic objects such as jewelry or metal clips;
* Women of childbearing age who are seeking to become pregnant, who are breastfeeding, or who suspect they may be pregnant;
* Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions;
* Any greater than normal potential for cardiac arrest

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Wave-CAIPI validation | 2 years
  The outcome measure for this project will be that the rapid scan from Wave-CAIPI can provide equivalent diagnostic quality to that of standard clinical acquisitions which is performed at much slower speed. This will be assess using visual qualitative assessment by experienced radiologists on the project.

CONTACTS AND LOCATIONS:
Overall Officials: Kawin Setsompop, PhD, Principal Investigator — Boston Children Hospital/ Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor- Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor- Investigator or designee].